CLINICAL TRIAL: NCT05812443
Title: Assessment of Sleep Quality and Mental Health After Using Meditation: a Randomized Controlled Trial
Brief Title: Assessment of Sleep Quality and Mental Health After Using Meditation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Rubens Lene Carvalho Tavares, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE: 60582522.5.0000.5149
Record Dates: First submitted 2023-03-17; First posted 2023-04-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Insomnia; Insomnia Chronic; Insomnia Disorder; Sleep Disorder; Anxiety Disorders; Stress Disorder; Depressive Disorder; Quality of Life; Complementary Therapy; Spirituality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Anxiety Disorders; Stress Disorders, Traumatic; Depressive Disorder | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shabad Kriya Meditation (Experimental): 87 participants (intervention group) will be trained to perform Shabad Kriya meditation for 30 minutes, daily, before going to sleep, for 8 weeks
  Interventions: Other: Shabad Kriya Meditation
- Relaxing reading (Active Comparator): 87 participants (control group) will perform relaxing reading for 30 minutes, daily, before going to sleep, for 8 weeks
  Interventions: Other: Relaxing reading

INTERVENTIONS:
Other: Shabad Kriya Meditation — The Shabad Krya meditation technique, used in Kundalini Yoga, will be performed by the participants of this intervention group for 8 consecutive weeks, for 30 minutes, before going to sleep. This group will be trained by a Kundalini Yoga teacher with extensive experience in Shabad Krya meditation. The evaluation of Sleep Quality, Mental Health and Spirituality parameters will be measured through specific questionnaires, shortly after the end of the eighth week of intervention, and also one month and three months after the end of the intervention.
  Other Names: Meditation
  Arms: Shabad Kriya Meditation
Other: Relaxing reading — Relaxing reading will be performed by the participants of this control group for 8 consecutive weeks, for 30 minutes, before going to sleep. The evaluation of Sleep Quality, Mental Health and Spirituality parameters will be measured through specific questionnaires, shortly after the end of the eighth week of intervention, and also one month and three months after the end of the intervention.
  Arms: Relaxing reading

SUMMARY:
This is a randomized controlled trial that intends to verify the effectiveness of the daily practice of meditation before going to sleep for the improvement of sleep, stress, mental health and quality of life of people with sleep problems.

DETAILED DESCRIPTION:
Participants selected for this clinical trial will be randomized into two groups: group 1 (intervention), with 87 participants undergoing 30 minutes of Shabad Kriya meditation before going to sleep, and group 2 (control), with 87 participants who will perform 30 minutes of relaxing reading before going to sleep. In addition, participants will complete the demographic data form; a sleep quality diary; and the scales: Pittsburgh Sleep Quality Index (PSQI), Perceived Stress Scale (PBS), Five Facets of Mindfulness (FFMQ), Daily Spiritual Experiences (DSES), Functional Assessment of Chronic Illness Therapy - Wellness Scale Spiritual (FACIT- 12), Duke Religiosity Index (DUREL), Quality of Life - Brief Mode (WHOQOL-Bref) and the Depression, Anxiety and Stress Scale (DASS 21). The study is open to the general community, and those interested are screened through the "Insomnia Severity Index" and questionnaires about health conditions. For conducting and guiding the intervention and completing the research instruments, online meetings will be held with the participants. The sleep quality diary will be completed for fourteen days before the start of the intervention (Baseline). Data collection will be carried out with online Google Forms questionnaires, sent through links in digital media, such as messages or emails, or made available in printed form. The main outcome measure will be sleep efficiency calculated using data from the sleep diary. Data from participants with ISI greater than or equal to 10 will be compared before and after the intervention. Additionally, data analysis of participants with ISI above or greater than 8 will be performed. At the end of the eighth week of the intervention (Shabad Kriya meditation or Relaxing reading), as well as one month after the end of the intervention, and three months after the end of the intervention, the participants will again fill in the questionnaires described above, for statistical comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of insomnia (Insomnia Severity Index between 8-28)

Exclusion Criteria:

* Major medical or psychiatric problems
* Who has used sleeping pills or sleep-disrupting medications in the last 30 days prior to participating in the study
* Who will need to use sleeping pills or sleep-disrupting medications during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mean Sleep Efficiency Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  Sleep efficiency is calculated as the number of hours asleep divided by the number of hours in bed with the intention to sleep. Sleep efficiency will be calculated from online sleep diaries that will be completed by participants in this study at baseline (T1), immediately after after 8 weeks of intervention (T2), 1 month (T3) and 3 months (T4) after intervention. Sleep efficiency is calculated using sleep parameters extracted from these diaries as sleep onset latency (SOL), total sleep time (TST), total wake time (TWT), Wake After Sleep Onset (WASO).

SECONDARY OUTCOMES:
Self-Reported Quality of Life Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  Self-reported quality of life will be measured at baseline (T1), immediately after after 8 weeks of intervention (T2), 1 month (T3) and 3 months (T4) after intervention using the Quality of Life - Brief Mode of World Health Organization (WHOQOL-Bref), a short 26-question version validated questionnaire. The WHOQOL-Bref provides a quality of life measure with four domain scores. Each item is weighted on a 0-5 interval scale. The WHOQOL-BREF score is then calculated according to the method described by the WHO, by totaling the 4 domain scores (physical health; psychological health; social relationships; and environment). The calculation method of the scores in a certain domain is: (summation of the scores in each domain) x 4 / (number of items in a category). The adjusted scores of each domain are as low as 4 points and as high as 20 points. The overall score ranges from 16 to 80, where higher scores denote a higher life quality.
Depression Anxiety Stress Scale (DASS)-21 Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  Change in Depression, Anxiety, and Stress will be measured using the Depression, Anxiety and Stress Scales short form (DASS-21). Each of the 21 items has a minimum value of 0 and a maximum value of 3, and summed to yield independent depression, anxiety, and stress scores. Higher scores indicate severe psychological distress.
Duke University Religion Index (DUREL) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Duke University Religion Index (DUREL) is a five-item measure of religious involvement. The instrument assesses the three major dimensions of religiosity that were identified during a consensus meeting sponsored by the National Institute on Aging (organizational religious activity, non-organizational religious activity, and intrinsic religiosity). The DUREL measures each of these dimensions by a separate "subscale". The DUREL has been used in many published studies conducted throughout the world and is available in many validated different languages questionnaires.
Insomnia Severity Index (ISI) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  Insomnia Severity Index (ISI) will be used to assess insomnia-related complaints. It is a short and easy self-applied scale with 7 items scored from 0 to 4, with a total score varying from 0 to 28. The total score is interpreted as follows: absence of insomnia (0-7); sub-threshold insomnia (8-14); moderate insomnia (15-21); and severe insomnia involvement. Patients are considered to be with no symptoms of insomnia if the ISI score is lower then 8. Data from participants with ISI greater than or equal to 10 will be compared before and after the intervention. Additionally, data analysis of participants with ISI above or greater than 8 will be performed.
Pittsburgh Sleep Quality Index (PSQI) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Pittsburgh Sleep Quality Index (PSQI) is a questionnaire that assesses sleep quality and disturbances over a 1-month period. Sleep quality will be measured by the Pittsburgh Sleep Quality Index. The PSQI has seven components, with a global PSQI score > 5 is indicative of poor sleep quality.
The Perceived Stress Scale (PSS) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Perceived Stress Scale (PSS) is a five-point Likert-type scale and consists of 14 items. Participants rate each item on a scale ranging from "Never (0)" to "Very often (4)". Seven of the items with positive statements are scored in reverse. As the scores obtained from the scale increase, the perceived stress level of the person increases. PSS-14 scores range from 0 to 56, with 0-35 point range indicating normal stress level, 35-56 point range indicating that the individual is under stress.
Functional Assessment of Chronic Illness Therapy (FACIT-Sp-12) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp-12) will be used to assess spiritual well-being and comprises 12 items, each rated on a 5-point scale by the respondent. The first eight items constitute the meaning/peace factor, and the last four items constituted the faith factor. The FACIT-SP-12 questionnaire assesses a sense of meaning, peace, and comfort and strength derived from faith. The FACIT-SP-12 has a 5-point Likert-type scale format. Total scores range from 0 to 48 with higher scores indicating higher levels of spiritual well-being.
Daily spiritual experiences scale (DSES) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Daily spiritual experiences scale (DSES) will be used to assess ordinary experiences of connection with the transcendent in daily life. It includes constructs such as awe, gratitude, mercy, sense of connection with the transcendent and compassionate love. It also includes measures of awareness of discernment/inspiration and a sense of deep inner peace. The DSES is a 16-item self-report measure questionnaire, and higher scores are associated with higher life satisfaction and self-reported good health. The first 15 items are arranged on a Likert-type scale, with scores ranging from 1 (many times a day) to 6 (never or almost never). The item 16 is answered on a 4-point scale (from 1 = not at all to 4 = as close as possible). The score of item 16 is inverted to maintain the same direction as the other items. The total score is obtained by adding the scores of the 16 items, ranging from 16 to 94. Lower scores reflect a higher frequency of spiritual experiences
Five Facet Mindfulness Questionnaire (FFMQ-BR) Change | Baseline (T1), after 8 weeks of intervention (T2), 4 weeks after the end of the intervention (T3), and 12 weeks after the end of the intervention (T4)
  The Five Facet Mindfulness Questionnaire (FFMQ-BR) will be used to assess the characteristics of mindfulness. The FFMQ-BR is subdivided into five main evaluation factors (observation, description, non-judgment, non-reactivity and conscientious acting) evaluated in the situations addressed in each item, and each item is rated by the participant using a scale ranging from 1 to 5 points, where 1 represents "never or almost never" and 5 represents "always or almost always". The total score of the questionnaire will be calculated and this score will be compared before and after all intervention to assess whether the participants' level of attention has increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khalsa SBS, Goldstein MR. Treatment of chronic primary sleep onset insomnia with Kundalini yoga: a randomized controlled trial with active sleep hygiene comparison. J Clin Sleep Med. 2021 Sep 1;17(9):1841-1852. doi: 10.5664/jcsm.9320. PMID 33928908
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Lin CY, Saffari M, Koenig HG, Pakpour AH. Effects of religiosity and religious coping on medication adherence and quality of life among people with epilepsy. Epilepsy Behav. 2018 Jan;78:45-51. doi: 10.1016/j.yebeh.2017.10.008. Epub 2017 Nov 22. PMID 29175219
- See also: Cultural adaptation and validation of the Underwood's Daily Spiritual Experience Scale - Brazilian version — https://doi.org/10.1590/S0080-62342012000700015